CLINICAL TRIAL: NCT01702649
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Ascending Single- and Multiple-Dose Study of the Safety, Tolerability, Pharmacokinetics of Intravenous RPX2003 in Healthy Adult Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics of Intravenous RPX2003 (Biapenem) in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rempex Pharmaceuticals (a wholly owned subsidiary of The Medicines Company) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rempex 401
Record Dates: First submitted 2012-09-25; First posted 2012-10-08 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Healthy Volunteers; Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — biapenem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- RPX2003 (Biapenem) (Experimental): Single and multiple dose of RPX2003 (Biapenem).
  Interventions: Drug: RPX2003 (Biapenem)
- Normal Saline (Placebo Comparator): Single and multiple doses of normal saline.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RPX2003 (Biapenem) — Six (6) cohorts of 3 active or 8 subjects of 6 active are planned for evaluation.
  Single dose followed by multiple dose, three times a day.
  Arms: RPX2003 (Biapenem)
Drug: Placebo — Six (6) cohorts of 1 placebo or 8 subjects of 2 placebo are planned for evaluation.
  Single dose followed by multiple dose, three times a day.
  Arms: Normal Saline

SUMMARY:
RPX2003 (biapenem) is being studied in combination with a beta-lactamase inhibitor to treat bacterial infections, including those due to multi-drug resistant bacteria.

DETAILED DESCRIPTION:
The worldwide spread of resistance to antibiotics among Gram-negative bacteria, particularly members of the ESKAPE group of pathogens, has resulted in a crisis in the treatment of hospital acquired infections. In particular, the recent dissemination of a serine carbapenemase (e.g., KPC) in Enterobacteriaceae in US hospitals now poses a considerable threat to the carbapenems and other members of the beta-lactam class of antimicrobial agents.

Rempex is developing a fixed combination antibiotic of a carbapenem (RPX2003 or biapenem) plus a new beta-lactamase inhibitor (RPX7009) which has activity against serine beta-lactamases, including KPC. This Phase 1 study will assess the safety, tolerability and pharmacokinetics of biapenem, administered alone, in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and/or females, 18 to 55 years of age
* Body mass index (BMI) ≥ 18.5 and ≤ 29.9 (kg/m2) and weight between 55.0 and 100.0 kg (inclusive).
* Medically healthy with clinically insignificant screening results
* Non-tobacco/nicotine-containing product users for a minimum of 6 months prior to Day 1.
* Sexually abstinent or use acceptable methods of birth control

Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
* History or presence of alcoholism or drug abuse within the 2 years prior to Day 1.
* Hypersensitivity or idiosyncratic reaction to compounds related to the study drug (e.g. beta-lactam antibiotics such as penicillins, carbapenems, etc).
* History of seizures (e.g., epilepsy).
* Use of any over-the-counter (OTC) medication, including herbal products and vitamins, within the 7 days prior to Day 1. Up to 2 grams per day of acetaminophen is allowed for acute events at the discretion of the PI.
* Blood donation or significant blood loss (i.e., > 500 mL) within 56 days prior to Day 1.
* Subjects who have any abnormalities on laboratory values at screening or check-in (Day -1).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Safety from baseline through the end of the study. | Study Day 1 to 13.
  Number of patients with adverse events; assessed by patient reporting, collection of vital signs, ECGs and absolute values and changes over time of hematology, chemistry and urinalysis.

SECONDARY OUTCOMES:
Composite of PK parameters RPX2003 & placebo following single dose administration. | Part 1A Study Day 1 to 3.
  plasma AUC0-t, AUC0-inf, Cmax, and Tmax.
Composite of PK parameters RPX2003 & placebo following multiple dose administration. | Part 1B Day 4 to 12
  plasma AUC0-t, AUC0-inf, Cmax, and Tmax.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Loutit, MBChB, Study Director — Sponsor GmbH
Locations (1):
- Celerion, Tempe, Arizona, United States